CLINICAL TRIAL: NCT02505061
Title: The Use of Modified ride-on Cars to Advance Mobility and Socialization in Young Children With Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: NSC102-2314-B-182-002
Record Dates: First submitted 2015-06-26; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-06

CONDITIONS: Children With Mobility Disabilities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Program (Experimental): The participant"s performance is indicative of the extent to which early power mobility training is feasible for both young infants and up to 3-year-old child with mobility Disabilities.Parents/caregivers and occupational therapists will be responsible for theHospital-based Program and Regular Therapy Program service respectively
  Interventions: Behavioral: Hospital-based Program; Behavioral: Regular Therapy Program

INTERVENTIONS:
Behavioral: Hospital-based Program — The research team will discuss with the clinical therapists who will provide training program in a hospital for 120 minutes/per session, 2 sessions/per week for a total of 9-week intervention. In addition, the research team will videotape the child"s natural play and driving performance at the hospital for 20 minutes/per session, 1 session/per week during the 9-week intervention phase. The treatment program of the two sessions will be preplanned and adjusted by the occupational therapist through clinical observation of participant's performance in the previous session. Training will still concentrate on building the concept of casual-effect on the switch and car motion, goal-oriented driving (e.g., driving 200 meters and reach for a toy or contact with a person), and upper limb use in functional tasks with driving in a hospital,discussed by the family, the treating therapist and the research team.
Behavioral: Regular Therapy Program — The regular therapy group will continue the regular therapy, including physical, occupational and speech therapy. The general propose of the training is to improve the developmental scales, mobility, socialization and upper limb use in functional tasks. The research team will videotape the child"s natural play and driving performance at the hospital for 20 minutes/per session, 1 session/per week during the 9-week intervention phase

SUMMARY:
The four purposes of this study are: 1) to examine the feasibility of providing children with disabilities to explore the environment with a modified ride-on car; 2) to quantify whether children with disabilities are able to have more social interactions with a ride-on car; 3) to examine the progression of socialization during the intervention and follow-up phases to determine which factors might influence the learning curve; 4) to compare the effectiveness of using the modified toy cars through the hospital-based program and regular therapy program after intervention and follow-up phases to determine the critical factors on increasing independent mobility and socialization, including motivation, treatment executor, treatment environment and play programs. It can provide guidelines for the future intervention.

Independent mobility is believed to be essential for perceptual-motor, cognition, language and social skill development. It is important to increase the independent mobility in children with disabilities and further enhance their development, especially motor and socialization. Assistive and power mobility devices allow children with disabilities to move independently within their environment and may increase the opportunities to explore and interact with people and environment . However, issues to consider before prescribing an assistive device include factors such as age, accessibly to community environments, cost, social acceptance of the device and the adaptability of the device to growth. This study is to use the customized, modified ride-on toy cars, to enhance the independent mobility, exploration and socialization through low-cost, family-centered approach. It will also improve family's understanding of children's capabilities, which improve their development. Investigators will recruit 60 children with who are between 1 to 3 years old and diagnosed as motor delay (>1.5 sd). They will be randomly assigned to one of the following two groups: hospital-based program group and regular therapy group.

The whole study duration will be 18 weeks, including 9-week intervention and 9-week follow-up; the total amount of treatment will be equal for two groups. The hospital-based program will be administered by the therapist and include 120 minutes/per session, 2 sessions/per week. In addition, the research team will visit the hospital once/per week to provide assessments. The regular therapy group will continue their regular therapy without any additional car driving training. The research team will visit them once/per week for the assessments. The assessments include behavior coding from the videotapes and the clinical assessments. The findings of this study will help to understand the feasibility and effectiveness of using the low-tech modified toy cars on advancing children's mobility and socialization. They can be used in the clinics and are a low cost alternative or addition to other mobility devices. They may provide a novel therapeutic tool to improve mobility, socialization and development.

DETAILED DESCRIPTION:
Children with mobility disabilities have more limited opportunities to explore their environment; therefore, they are considered to be at risk of secondary impairments, such as cognitive, spatial-perceptual, and social-emotional delay. Independent mobility is believed to be essential for perceptual-motor and social skills development. Self-produced locomotion is an organizer of psychological changes in typically developing infants/children, especially developmental changes in perceptions, social understanding, spatial cognitive, and emotions. Power mobility devices provide the potential for children with disabilities to move more independently and increase their exploration and interaction with the social and physical environment. Through the exploration, infants can detect the object and individual"s information that relates size, orientation, shape, substance to their perceptual and movement capabilities and interpersonal relationships. Logically, starting powered mobility as part of a comprehensive Early Intervention (EI) program within the first year of life should not only provide mobility but also reduce secondary impairments for children with disabilities. Although of increasing interest, there is very little empirical evidence of the effects or even feasibility of early power mobility training on development, particularly for mobility and socialization. A hallmark of daily life for the typically developing infants and toddlers is hours of mobility nested within exploration, socialization and object play in the home and community.Pediatric rehabilitation, through training and assistive technology (AT), seeks to provide children with disabilities with this same level of mobility, exploration and socialization. There are many basic barriers to achieving this high standard and no single AT or combination of AT can currently provide the level of mobility that children, families and therapists desire. For example, certain characteristics of the most common commercial pediatric power wheelchairs limit their use in the home and community spaces such as playgrounds. These limitations include price (e.g., typically $5000), size and weight (e.g., typically >150 lbs), transportation requirements (e.g., van or truck), maintenance and aesthetics and social acceptance. The most obvious limitation for including power mobility in EI programs is the complete lack of readily available power chairs for children younger than 2-3 years of age, the period when mobility is rapidly developing for typically developing children. Experimental power mobility devices have the potential to address some of these limitations such as size, weight and infant use. Unfortunately these are likely years from commercial availability. Furthermore, power wheelchairs have historically been designed to address a limited set of goals related to mobility with minimal consideration of socialization. Investigators believe there is a need for readily available mobility options for immediate use by very young children and their families that address some of the above limitations while expanding the role of power devices past simply mobility and into socialization. The general purpose of this study is to determine the feasibility of using a "ride-on toy car" as an early option for power mobility. Furthermore, this study will examine the effects of using a toy car to advance mobility and socialization in the early development. The use of modified ride-on toy cars may provide a readily available, convenient and fun way for families, therapists and early educators to help young children improve their mobility starting within the first years of life. There are four strengths of using ride-on toy cars for mobility. First, the cost is comparable or less than most mobility devices. Second, most are relatively lightweight, small and easily transported in contrast to power chairs. Third, the child-friendly, colorful toy designs are more acceptable to adults and children and likely seen as simply a toy. This may be an important aspect for clinicians wanting to start early power mobility training with families hesitant to discuss powered chair options. Fourth, because toy cars are simple electromachanical devices, they can be modified quickly and easily to match the child's current and/or future abilities and goals. Ride-on cars provide fun and mobility for typically developing children and have serious potential to be a power mobility option for children with disabilities. Investigators have recently published a technical report outing the basic components and exemplar modifications. Our pilot study has also shown positive effects on increased socialization in a 2-year old child with severe cerebral palsy. No studies have been published on the effectiveness or even the feasibility of including these cars with any pediatric population. Thus basic questions such as sitting tolerance, basic driving ability and interest in using the car for socialization have not been addressed prior to wide spread clinical use. The long term effects of using this mobility device on mobility and socialization also remain a question for the researchers and clinicians. In addition, little is known about the learning curve of using the power mobility device to improve mobility and socialization, e.g., at what point in time (maximal) effects are reached. Up to now, most of the studies have focused on the end results of increased amount of independent mobility in daily life. It is still unknown whether optimal (maximal) effects are being reached at all and which factors (e.g., training environment, training executor) might influence the learning curve as well as the retention of treatment effects in the long term. In the study by Tieman et al. (2004), they suggested that therapists should examine children's performances in the settings that are important to their daily life. Examining performance in everyday settings enables the therapists not only to observe the child's ability, but also to assess environmental features that either facilitate or hinder mobility. Our study will focus on providing intervention and exploratory assessments in the home or a clinical setting. This information is essential for making future decisions on whether interventions should focus on the child"s motor ability in a therapeutic environment from the therapist's perspective, or adaptation of the natural environment for the caregiver's application. In this study, investigators will modify ride-on toy cars for children with disabilities for use in the clinical settings as part of a 18-week power mobility training program. Investigators focus on four basic questions. Specifically, can investigators: 1) select and modify toy cars such that children with motor impairments enjoy sitting and driving, 2) select a set of dependent measures that quantify whether the children increase their independent mobility and socialization; 3) determine the factors that influence the learning curve of independent mobility and socialization during intervention and follow-up phases; 4) conduct a hospital-based training program that results in a high level of fun for the child and compliance by the family and therapists. If our results are generally positive and show significant differences between different programs, then future randomized controlled trial studies could further quantify the effectiveness and the feasibility with different treatment intensity and various pediatric populations.

Evidence supported that independent mobility might improve different skills for children with mobility impairments, including spatial awareness skills, eye-hand coordination, visual perceptual skills, spontaneous vocalizations, initiation of contact with others,motivation to explore and an increased ability to interact meaningfully with peers. Although the mobility devices are considered to be used to compensate for disabilities causing difficulties with the accomplishment of daily activities and social roles, the current standard of clinical practice in the United States for power wheelchair training is that children must demonstrate certain prerequisite abilities before they are eligible. As a result, power mobility training, based on readiness, if offered clinically to children between 2 and 6 years old, with 3 years being the average age of the youngest child being recommended for a power wheelchair.However, several studies have demonstrated that early power mobility training is feasible, even for the children who may be categorized as in a "not-ready" group based on their age, motor or cognitive abilities. These children had various types of disabilities which limited their self produced locomotion. Most of them were younger than 3 years of age and the youngest one was only 7-month-old. The early power mobility training allowed these young children with mobility impairments move independently and have positive impacts on overall development. The investigators reported increased vocalizations, increased arm and hand movements, greater motivation to explore,increased self-confidence and curiosity and positive effects on family life in these children. Power mobility devices can not only be designed to compensate children's impairments for independent mobility, but also be used as a novel, training device to address socialization, body functions, activity and participation goals. Combined with a family centered (e.g., coaching of parents), functional approach which aims to promote better functioning in the context of daily life settings (e.g., home environment), early power mobility training can help to enhance development and improve social participation in children's daily life. Current power wheelchairs have limitations that limit their functional use in the community. These include their size, weight, cost, accessibility, ease of transportation, maintenance requirements, adaptability to the body growth and social acceptance. Experimental devices have the potential to address some limitations such as size, weight and cost but may be years from commercial availability. Providing a new option of device for early power mobility which addresses these environmental limitations is necessary. Furthermore, this device can also be used to focus on the three ICF levels as a training tool. For example, our technique report of modifying ride-on toy cars as power mobility devices introduces an alternative way to provide early power mobility training. Compared to traditional pediatric power wheelchairs, the strengths of modified toy cars include less cost, more accessibility to community environments, better aesthetic and adjustability. Moreover, a modified toy car is unlike a powered wheelchairs which is a medical device and typically focuses on activity and participation levels of ICF. Various permanent and temporary modifications of a toy car allow clinicians to address one or more ICF levels. For example, more trunk support may help a child to reach the steering wheel and grasp toys during car movement to address an ICF activity goal. By lessening the trunk support modifications in combination with a simple steering system (e.g., a push-button switch), clinicians can provide the child with a more challenging, dynamic postural control during driving to address an ICF body functions and structure goal. The child-friendly frame of the toy car can motivate a child's exploratory behaviors and may have positive impacts on family's and/or other people's perceptions of a child's capabilities. These strengths of a ride on toy car make it become the appropriate candidate for the family and therapists to improve early independent mobility and socialization for children with mobility disabilities.

The specific aims of this study are: 1) to examine the feasibility of providing children with disabilities to explore the environment with a modified ride-on car; 2) to quantify whether children with disabilities are able to have more social interactions with a ride-on car; 3) to examine the progression of socialization to determine which factors might influence the learning curve during intervention and follow-up phases; 4) to compare the effectiveness of using the modified toy cars through the hospital-based program and regular therapy program to determine the critical factors on increasing independent mobility and socialization after intervention and follow-up phases, including motivation, treatment executor, treatment environment and play programs. Through the comparison of Car Play (i.e., play with the use of toy cars) and Natural Play (i.e., play without the use of toy cars), investigators hypothesize that children with disabilities are able to learn how to drive the modified toy cars in the hospital-based group. They will have increased socialization (i.e.,self-initiated contacts, vocalizations, positive facial expressions) when driving the cars than the regular therapy program, i.e., control group.

Study Design: A pretest-posttest control group design was applied. Two groups were involved in this project: hospital based program, and regular therapy program. The participants were randomly assigned to one of the two groups by using the well-sealed, opaque envelopes when they are recruited in the study. Once the participants were recruited in the study, the research team modified a toy car based on each participant's capabilities during this pre-intervention phase (the first two or three weeks before intervention starts), e.g., seat and steering wheel modifications. The study duration for each participant was 18 weeks, including 9-week intervention and 9-week follow-up.

Participantsin the study were 60 infants or preschool children ages 12 months to 36 months with motor delays (sd > 1.5). The age group of infants/preschool children was selected based on the previous studies on early power mobility training in infants and preschool children. Power mobility training was typically offered to children between two and six years of age, with three years being the average age of the youngest child being recommended for a powered chair. However, studies showed that early power mobility training was feasible for 7-month-old infants and 18-month-old children with mobility disabilities.

Recruitment: The children were recruited from self-referrals, health care practitioners, or the hospitals in Taipei and Taoyuan, Taiwan where children with motor delays (>1.5 sd) were receiving outpatient rehabilitation. The research team initially posted flyers describing the study at clinical settings and contacted the therapists in the clinical settings to introduce the goals,criteria and general procedure of the study. Parents/guardians obtained information about the study through the flyers and their therapists. Parents/guardians, who were interested and whose children met the criteria of diagnosis, age, capability determined by the doctor and their therapists, were given contact information for the investigator. After receiving contact information, the research team contacted the parents/guardian and/or therapists for scheduling a date of further testing by the research team at the hospital. When the research team contacted the parents, study was explained and parents received a letter detailing the procedure and given an opportunity to ask questions. Parents/guardians signed this informed consent form at the time of the first visit.

Procedure: Before the pre-intervention assessments, the research team modified the car's seat and acceleration to the hand switch-driven, which allowed the car to be drivable for the child who met the inclusion criteria. Each child had a customized ride-on toy car in a hospital. After modifications, they received pre-intervention assessments, including behavioral videotaping and developmental assessments. The developmental assessments occurred at the first and last week of the 9-week intervention, and the end of the 9-week follow-up phase. A therapist who did not involve in the intervention and was blinded to the study purpose completed all the developmental tests. The driving and socialization behaviors were videotaped by the research team for 20 minutes/per session, one session/per week before, during and after the intervention phase at the child house or a hospital. All videotapes were coded by two independent coders, who were undergraduate students. Prior to making their ratings, the coder was instructed as to coding procedures by the PI, but he/she was not informed about the group assignment and the purpose of the study. Cohen's kappa coefficient was calculated between the two independent raters to establish good reliability before formal coding.

Intervention: Parents/caregivers and occupational therapists were responsible for the hospital-based rehabilitation service. For the hospital-based program, the research team discussed with the clinical therapists who provided training program in a hospital for 120 minutes/per session, 2 sessions/per week for a total of 9-week intervention. In addition, the research team videotaped the child's natural play and driving performance at the hospital for 20 minutes/per session, 1 session/per week during the 9-week intervention phase. The treatment program of the two sessions was pre-planned and adjusted by the occupational therapist through clinical observation of participant's performance in the previous session. Training concentrated on building the concept of casual-effect on the switch and car motion, goal-oriented driving (e.g., driving 200 meters and reach for a toy or contact with a person), and upper limb use in functional tasks with driving in a hospital,discussed by the family, the treating therapist and the research team.

Regular Therapy Program: The regular therapy group continued the regular therapy, including physical, occupational and speech therapy. The general propose of the training was to improve the developmental scales, mobility, socialization and upper limb use in functional tasks. The research team videotaped the child's natural play and driving performance at the hospital for 20 minutes/per session, 1 session/per week during the 9-week intervention phase.

Follow-up: This period focused on the 9 weeks follow-up after receiving a treatment program. No treatment program was delivered to the participants. The research team still videotaped the child's natural play and driving performance at the hospital for 20 minutes/per session, 1 session/per week during the 9-week follow-up phase.

Instrument and Procedure: Each participant received pre-intervention assessments, including behavioral videotaping and developmental assessments. Behavioral coding involved the mobility/driving performance during the 10-minute Car Play and socialization during the whole 20-minute Play (i.e., 10-minute Natural Play and 10-minute Car Play). The developmental assessments occurred at the first and last week of 9-week intervention, and the end of the 9-week follow-up phase, including the Pediatric Evaluation of Disability Inventory (PEDI), the Bayley Scales of Development, and Parenting Stress Index (PSI). Necessary materials include two video cameras, a parent log and a customized ride-on car.

Data Reduction and Analysis: All videotapes will be coded by two independent coders, who are undergraduate students. Prior to making their ratings, the coder is instructed as to coding procedures, but he/she is not informed about the group assignment and the purpose of the study.

Mobility Measures: The following measures were obtained via video coding the 10-minute Car Play during pre-intervention, intervention and post-intervention phases to determine the feasibility of learning to drive the car:

1. Driving Categories (time in seconds)

   a. Independent Mobility: When the child independently drives the car preceded by an independent switch contact without an adult's assistance. b. Assisted Mobility: When an adult puts the child"s hand on the switch but he independently pushes the switch to begin driving. c. Caregiver Mobility: When the child drove with an adult"s hand directly on top of his hand.
2. Visual Attention to Switch: The frequency (number of times) that the child looked at the switch during the 10-minute driving.
3. Stopping Categories (number of times divided by total times goal was presented) a. Independent Stop: When the child independently moves his hand off the switch and makes the car stop within one car length of the goal location. b. Stops with Verbal Cues: When the child moves his hand off the switch as the car arrives the goal only after verbal cues given from an adult. c. Stops with Tactile Contacts: When the child moves his hand off the switch as the car arrives the goal only after tactile cues (e.g., touching his hand or moving his hand off the switch) given from an adult

Socialization Measures: To examine the impact of independent mobility on the socialization during the 10- minute Natural Play and 10-minute Car Play, the following measures will be obtained via coding video footage during pre-intervention, intervention and post-intervention:

1. Reaching for toy/person: The frequency (number of times) that the child initially extends arms to the play toy/interacting person.
2. Initiation of contact with others: peer-directed or adult-directed: Target child-initiated contacts with others are counted whenever two conditions are met: (a) the target child initiates the contact with another individual without any observable prompting or initiating behavior on the part of another person and (b) the target child independently vocalizes (with either comprehensible words or other vocalizations, including shouting,laughing, grunting, etc.) or physically points to, touches, or indicates that he or she wants something from another individual. Target child-initiated contacts and vocalizations are divided into two categories: (i) peer-directed and (ii) adult-directed.
3. Other initiated contacts: contact by peers or by adults: Peer-initiated contacts are defined as any child initiating any type of contact with the target child (e.g., talking to the child, touching the child or a mobility device the child is using, giving a toy or item to the child,taking a toy or item away from the child). Adult-initiated contacts with the target child are: (a) carrying, moving, or otherwise touching the child or the device in which the child is seated (e.g., swing, wheelchair, toy car); (b) taking a toy or item away from the child
4. Facial Expression: The frequency (number of times) of both positive and negative facial expressions appeared during interaction. Positive was determined to include smiling and laughing. Negative was determined to include discomfort, crying and unhappy facial expression.
5. Vocalization/Gesture: The frequency (number of times) that the child vocalizes/gestures to a play toy or person, including grunting, shouting, vowel-type sounds (e.g., ee, i, ah, oo u).

Repeated measure one way ANOVA was used to compare the mean difference of using a toy car for mobility, socialization and development before and after the intervention, and the follow-up. One way ANOVA was used to compare the mean difference of all developmental tests (mobility, socialization, motor, cognition) between two groups before and after the intervention and the end of follow-up phase. To analyze the learning curve, the results of socialization will be individually examined for each participant in two groups. The instant of the maximum training effect will be defined as the moment the top of the learning curve is reached. This top will be independently determined by two coders through visual examination of the absolute values. Subsequently, the data set will be split in children that have reached a maximum effect within the 9 weeks intervention period and those who have not. These two groups will then be compared with regard to demographic (age, gender) and clinical (manual ability classification system-MACS, gross motor function classification system-GMFCS) characteristics (using X2-test for dichotomous variables and Mann-Whitney U test/or t-test for the MACS and GMFCS depending on the normality of data).

ELIGIBILITY:
Inclusion Criteria:

1. motor delays (sd>1.5) resulting in motor impairments that prevented functional independent mobility, such as rolling, crawling, walking;
2. aged between 12 months to 36 months old;
3. able to tolerate sitting with support for 30 minutes;
4. able to reach the objects with either one or two hands;
5. consent of the parents to agree to the testing procedures and participate in the training program at their own house or at the hospital.

Exclusion Criteria:

1. children with severe sensory impairments such as blindness, deafness,
2. parents/caregivers are not able to make a time commitment for the training phase.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in General Mobility and Social Development at 9 weeks and 18 weeks as assessed by the Pediatric Evaluation of Disability Inventory (PEDI) | Assessment occurred 3 times during the whole study, including the first and last week of the 9-week intervention, and the end of the 9-week follow-up phase.
  PEDI is a set of tests for children from 8 months to 6 years old. The PEDI quantified self-care, mobility, and social functions. The PEDI is especially useful for tracking changes in functional skills.
Mobility/Driving Performance as assessed by the coding behaviors from the videotaping | The driving behaviors were followed for the duration of implementing the intervention program at the hospital, an expected average of 9 weeks.
  The driving behaviors were coded from each 10-minute Car Play session: a) amount of time moving/total time, b) frequency, time and duration of parental assistance (physical and/or vocal), c) number of successful "directional driving trials". In each of 10 trials, the child is asked to drive 5 feet to the parent or researcher. He/she is given 30 seconds to complete the distance and make a stop at the goal.
Socialization as assessed by the coding behaviors from the videotaping | The socialization behaviors were followed for the duration of implementing the intervention program at the hospital, an expected average of 9 weeks.
  The frequency and duration related to socialization were coded during the whole 20-minute Play, including 10-minute Natural Play and 10-minute Car Play: physical contacts, initiation of contact with others, other initiated contacts, facial expressions, vocalizations/gestures and mutual play events (ex. sharing a toy).

SECONDARY OUTCOMES:
Change from baseline in General Development at 9 weeks and 18 weeks as assessed by The Bayley Scales of Development | It was administered a total of 3 times during the whole study, including the beginning and end of the 9-week intervention, and the end of the 9-week follow up.
  The Bayley Scales of Development is an internationally recognized set of developmental tests that involve play and parental questionnaires. The Bayley has subsets of tests for motor (fine and gross), language (receptive and expressive), and cognitive development, ages from 0-3 years old.
Change from baseline in Parents' Perceptions at 9 weeks and 18 weeks as assessed by Parenting Stress Index (PSI) | It was administered a total of 3 times during the whole study, including the beginning and end of the 9-week intervention, and the end of the 9-week follow up.
  PSI is a tool that was designed to measure the overall level of parenting stress experienced by parents of children between the ages of one month and twelve years.